CLINICAL TRIAL: NCT04663100
Title: Oral Adherence in Hematological Oncology Agents and Impact on Comorbid Therapy Adherence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee (Other)
Collaborators: Vanderbilt University Medical Center (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-0839
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Chronic Myeloid Leukemia; Chronic Lymphocytic Leukemia; Multiple Myeloma; Multiple Chronic Conditions
Keywords: adherence; leukemia; anticancer agents; chronic disease management; pharmacy practice; hematological malignancy
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Multiple Chronic Conditions; Leukemia; Hematologic Neoplasms | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacist Coordinated care Oncology Model (Experimental): The Pharmacist Coordinated care Oncology Model includes patient self-reported symptoms and medication adherence, comprehensive medication review(s) and intentional communication between oncology and community pharmacists.
  Interventions: Other: Patient-reported outcome measure; Other: Comprehensive Medication Review; Other: Pharmacist communication

INTERVENTIONS:
Other: Patient-reported outcome measure — Participants will complete a patient-reported outcome measure for their oral anticancer agent at two timepoints over 2 months, to assess patient symptoms and adherence to their oral anticancer agent.
Other: Comprehensive Medication Review — Following the first patient-reported outcome measure, participants will be contacted by the community pharmacist for a Comprehensive Medication Review (CMR) for their chronic medications. A follow-up CMR will take place after the second patient-reported outcome measure.
Other: Pharmacist communication — Throughout the study, the oncology and community pharmacists will communicate about medications through the electronic medical record.

SUMMARY:
The objective of this study is to improve medication, symptom, and disease management of patients with hematological malignancies and multiple chronic conditions (2 or more conditions in addition to cancer) through care coordination between pharmacists working in oncology practices and those working in primary care or community practices (Pharmacists Coordinated care Oncology Model [PCOM]).

This is a pilot study in which the investigators will examine the association between outcome measures, but the study design and sample size are insufficient to quantify the impact of OAA initiation or OAA adherence on adherence to chronic medications. This pilot study and data analyses are being done in preparation for a larger, controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Receiving cancer care at Vanderbilt University Medical Center
* Diagnosis of chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), chronic myeloid leukemia (CML), or multiple myeloma (MM)
* Initiating an oral anticancer agent, either for the first time or a change from previous oral agent
* Diagnosis of 2 chronic conditions, including at least one of the following: diabetes, hypertension, hyperlipidemia, congestive heart failure, depression/anxiety, gastroesophageal reflux disease, and/or chronic obstructive pulmonary disease
* Patients taking at least two chronic medications, including at least one medication for one of the conditions listed above.
* Willing and able to sign informed consent.

Exclusion Criteria:

* Cannot communicate in English
* Concurrent diagnosis of type 1 diabetes or human immunodeficiency virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Oral anticancer agent adherence by proportion of days covered (PDC) | Up to 6 months post-initiation
  PDC is a common medication adherence metric, and assesses the ratio of number of days the patient is supplied with oral anticancer agent, from the time of initiation until 6 months later, to the total number of days during that period. Data from the electronic medical record for dose changes will be aligned with the refill data to calculate a dose-adjusted PDC.
Chronic disease medication adherence | 6 months pre- and post-initiation of the oral anticancer agent
  PDCs for medications for select chronic diseases will be calculated for the 6 months before and after oral anticancer agent initiation

SECONDARY OUTCOMES:
Patient-reported outcome measure completion | Approximately 42 days after oral anticancer agent initiation
  The oncology-specific patient-reported outcome measure is to be completed at 2 and 6 weeks after oral anticancer agent initiation. This measure assesses the percent of patients who complete this tool at both time points.
Comprehensive Medication Review (CMR) completion | Approximately 50 days after oral anticancer agent initiation
  Proportion of enrolled subjects completing the initial and follow-up CMRs with the community pharmacist
Oncology pharmacist review of patient-reported outcome measure | Approximately 44 days after oral anticancer agent initiation
  The patient-reported outcome measure is scored within one day after it is completed by the subject and is routed to the oncology pharmacist to review the results. The number of measures that are reviewed within 1 day of receipt will be assessed at 2 weeks and at 6 weeks.
Percent of Comprehensive Medication Reviews (CMRs) where note was routed to oncology pharmacist | Approximately 43 days after oral anticancer agent initiation
  The number of CMRs where note was routed to oncology pharmacist out of total number of completed CMRs, assessed at 2 weeks and at 6 weeks.
Proportion of Comprehensive Medication Reviews (CMRs) reviewed by the oncology pharmacist | Approximately 44 days after oral anticancer agent initiation
  The number of CMR notes reviewed by the oncology pharmacist out of the total number of completed CMRs, assessed at 2 weeks and at 6 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No